CLINICAL TRIAL: NCT04702737
Title: A Phase 1b Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of Delta-like Protein 3 Half-life Extended Bispecific T-cell Engager AMG 757 in Subjects With De Novo or Treatment Emergent Neuroendocrine Prostate Cancer
Brief Title: A Study of AMG 757 in Participants With Neuroendocrine Prostate Cancer
Acronym: DeLLpro-300
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20200040
Expanded Access: NCT06064500 (Approved for marketing)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Neuroendocrine Prostate Cancer
Keywords: De novo or treatment emergent neuroendocrine prostate cancer; Non-canonical Notch ligand
MeSH Terms: interventions — AMG 757

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Exploration (Experimental): The maximum tolerated dose (MTD) will be estimated using isotonic regression (Ji et al, 2010). The recommended phase 2 dose (RP2D) may be identified based on emerging safety data prior to reaching an MTD.
  Interventions: Drug: Tarlatamab
- Part 2: Dose Expansion (Experimental): Participants will receive the RP2D/MTD identified in Part 1 (dose exploration) of the study.
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Tarlatamab — Tarlatamab will be administered as an intravenous (IV) infusion.
  Other Names: AMG 757

SUMMARY:
To evaluate the safety and tolerability of Tarlatamab and will determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria (Part 1: Dose Exploration and Part 2: Dose Expansion):

* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* Men aged ≥ 18 years at time of signing the informed consent.
* Metastatic de novo or treatment-emergent neuroendocrine prostate cancer (NEPC) defined by histology, immunohistochemistry, or genomic analyses of baseline tumor tissue (by local assessment) or circulating tumor DNA (ctDNA) (by local assessment) as per protocol
* At least 1 line of prior systemic treatment per protocol.
* Participants with treatment-emergent NEPC or de novo NEPC with histologic evidence of prostate cancer with neuroendocrine differentiation without a history of bilateral orchiectomy are required to remain on luteinizing hormone-releasing hormone (LHRH) analogue therapy during the course of protocol therapy
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 per Prostate Cancer Working Group 3 (PCWG3) modifications
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Participants with treated brain metastases are eligible provided they meet defined criteria
* Adequate organ function as defined in protocol

Exclusion Criteria (Part 1: Dose Exploration and Part 2: Dose Expansion):

* History of other malignancy within the past 2 years, with exceptions:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 2 years before enrollment and felt to be at low risk for recurrence by the treating physician
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated non-muscle invasive urothelial carcinoma
* History or presence of hematological malignancies unless curatively treated with no evidence of disease ≥ 2 years
* Untreated or symptomatic brain metastases and leptomeningeal disease
* Anti-tumor therapy within 28 days of study day 1; concurrent use of hormone deprivation therapy for hormone refractory prostate cancer is permitted; participants on a stable bisphosphonate or denosumab prior to study day 1 are eligible

Exceptions:

* Participants who received conventional chemotherapy are eligible if at least 14 days have elapsed and if all treatment-related toxicities have resolved to Grade ≤ 1
* Prior palliative radiotherapy must have been completed at least 7 days before the first dose of tarlatamab
* Participants who received androgen signaling inhibitor are eligible if at least 14 days have elapsed and if all treatment-related toxicity has been resolved to Grade ≤ 1

  * Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior study day 1
  * Active autoimmune disease requiring systemic treatment within the past 2 years
  * Known positive test for human immunodeficiency virus (HIV) or hepatitis
  * Unresolved toxicities from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 grade 0 or 1 (with the exception of alopecia or toxicities that are stable and well-controlled)
  * History of hypophysitis or pituitary dysfunction
  * Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
  * Participants on prior delta-like ligand 3 (DLL3)-targeted therapy may be eligible if discussed with Amgen Medical Monitor prior to enrollment
  * Evidence of severe acute respiratory syndrome coronavirus 2 (SARS-COV2) infection unless agreed upon with Medical Monitor and with no acute symptoms of coronavirus disease 2019 (COVID19) disease within 14 days prior to first dose of investigational product (counted from day of positive test for asymptomatic participants).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 41 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (21):
- United States (10):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of California at San Francisco Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Community Health Network MD Anderson Cancer Center - North, Indianapolis, Indiana
  - Washington University, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Austria (3):
  - Medizinische Universitaet Graz, Graz
  - Ordensklinikum Linz Elisabethinen, Linz
  - Landeskrankenhaus Salzburg, Salzburg
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Gustave Roussy, Villejuif, France
- Keio University Hospital, Shinjuku-ku, Tokyo, Japan
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia, Spain
- Royal Marsden Hospital, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Aggarwal R, Rottey S, Bernard-Tessier A, Mellado B, Kosaka T, Stadler WM, Horvath L, Greil R, O'Neil B, Siddiqui BA, Bauernhofer T, Bilen MA, Eskens F, Sandhu S, Shaw C, Ju CH, Decato BE, Yu B, Aparicio A. Safety and Efficacy of Tarlatamab in Patients with Neuroendocrine Prostate Cancer: Results from the Phase 1b DeLLpro-300 Study. Clin Cancer Res. 2025 Sep 15;31(18):3854-3863. doi: 10.1158/1078-0432.CCR-25-1211. PMID 40689871
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 41 participants were enrolled into this study in the United States, Australia, Austria, Belgium, France, Japan, Netherlands, and Spain between June 2021 and July 2024.
Pre-assignment Details: The planned Part 1 did not enrol participants. It was eliminated as pre-specified in the protocol due to sufficient data from Study 20160323 (NCT03319940) at the time of study initiation allowing the recommended phase 2 dose (RP2D) of tarlatamab to be determined for Part 2. Therefore no dose escalation occurred during the study.
Groups:
- Tarlatamab Dose Expansion: Participants received tarlatamab as a short term IV infusion Q2W in a 28 day cycle until disease progression. All participants received the same target dose of tarlatamab which was reached using a step-dosing approach including a run-in dose on day 1 of the first cycle.
Period: Overall Study
Arm/Group | Tarlatamab Dose Expansion
Started | 41
Participants Who Received Treatment | 40
Completed | 1
Not Completed | 40
Not completed — Decision by Sponsor | 1
Not completed — Withdrawal of Consent from Study | 3
Not completed — Lost to Follow-up | 1
Not completed — Death | 35

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who were enrolled and received at least 1 dose of tarlatamab.
Arm/Group | Tarlatamab Dose Expansion
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced One or More Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. A TEAE was defined as an AE starting on or after the first dose of tarlatamab, and up to and including 47 days after the last dose of tarlatamab excluding the events reported after End of Study date. Clinically significant changes from baseline in vital signs, 12-lead electrocardiograms (ECGs) and clinical laboratory tests were also reported as TEAEs.
Time Frame: Up to approximately 3 years
Population: Safety Analysis Set: all participants who were enrolled and received at least 1 dose of tarlatamab.
Measure: Count of Participants; unit: Participants
Arm/Group | Tarlatamab Dose Expansion
Number analyzed (Participants) | 40
Participants | 40

2. Primary Outcome: Number of Participants Who Experienced One or More Treatment-related Adverse Events (TRAE)
Description: A TRAE was defined as a TEAE that per investigator review had a reasonable possibility of being caused by tarlatamab. Clinically significant changes from baseline in vital signs, 12-lead ECGs and clinical laboratory tests were also reported as TEAEs.
Time Frame: Up to approximately 3 years
Population: Safety Analysis Set: all participants who were enrolled and received at least 1 dose of tarlatamab.
Measure: Count of Participants; unit: Participants
Arm/Group | Tarlatamab Dose Expansion
Number analyzed (Participants) | 40
Participants | 40

3. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as any qualifying toxicity that was at least possibly related to tarlatamab with an onset within the first 28 days following first dose with either of the following criteria:
  1. Grade 3 adverse event lasting more than 3 days (with the exception of fatigue and Grade 3 non-febrile neutropenia that improved to ≤ Grade 1 within 3 weeks including the use of growth factor support per neutropenia management guidelines);
  2. ≥ Grade 4 adverse event regardless of duration (with the exception of grade 4 non-febrile neutropenia lasting less than or equal to 7 days including the use of growth factor support per neutropenia management guidelines).
Time Frame: Up to 28 days
Population: DLT Analysis Set: all participants who were enrolled and received at least 1 dose of tarlatamab with an evaluable DLT endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Tarlatamab Dose Expansion
Number analyzed (Participants) | 30
Participants | 1

4. Secondary Outcome: Objective Response Rate (ORR)
Description: OR was assessed per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 with Prostate Cancer Working Group 3 (PCWG3) modifications. OR was defined as best overall response of partial response (PR) or complete response (CR) per RECIST 1.1, confirmed by an assessment at least 4 weeks later. Participants who did not experience a PR/CR or did not have any follow-up tumor assessments were regarded as non-responders. ORR was defined as the percentage of participants with a best overall response of confirmed CR or PR per RECIST 1.1. The percentage of participants with an OR was summarized along with the Clopper-Pearson (Clopper and Pearson, 1934) exact 95% confidence interval (CI). The result reported was evaluated by central reviewer assessment.
Time Frame: Up to approximately 3 years
Population: Evaluable by Central Reviewer Analysis Set: all participants who were enrolled, received at least 1 dose of tarlatamab, had measurable baseline disease per RECIST 1.1 with PCWG3 modifications as assessed by a central reviewer.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tarlatamab Dose Expansion
Number analyzed (Participants) | 25
percentage of participants | 12.0 [2.5 to 31.2]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of an initial objective response to the earlier of progressive disease or death for participants with an objective response per RECIST 1.1. DOR was assessed per RECIST 1.1 with PCWG3 modifications. The distribution of DOR was summarized using the Kaplan-Meier (KM) method with CI calculated using the Brookmeyer and Crowley (Brookmeyer and Crowley, 1982) method. The result reported was evaluated by central reviewer assessment.
Time Frame: Up to approximately 3 years
Population: Evaluable by Central Reviewer Analysis Set: all participants who were enrolled, received at least 1 dose of tarlatamab, had measurable baseline disease per RECIST 1.1 with PCWG3 modifications as assessed by a central reviewer. Only participants with a confirmed response have been included here.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tarlatamab Dose Expansion
Number analyzed (Participants) | 3
months | NA [NA to NA] — The median KM DOR and 95% confidence interval could not be estimated due to all responders being censored.

6. Secondary Outcome: Radiographic Progression-free Survival (PFS)
Description: Radiographic PFS was defined as the interval from the first dose of tarlatamab to the earlier of a radiographic progression or death from any cause. Radiographic PFS was assessed per RECIST 1.1 with PCWG3 modifications. The distribution of radiographic PFS was summarized using the KM method with CI calculated using the Brookmeyer and Crowley (Brookmeyer and Crowley, 1982) method. The result reported was evaluated by central reviewer assessment.
Time Frame: Up to approximately 3 years
Population: Safety Analysis Set: all participants who were enrolled and received at least 1 dose of tarlatamab. Censoring was at the last evaluable disease assessment date (tumor assessment or bone scan).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tarlatamab Dose Expansion
Number analyzed (Participants) | 40
months | 2.1 [1.8 to 3.8]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the start of treatment until event of death due to any cause. The distribution of OS was summarized using the KM method with CI calculated using the Brookmeyer and Crowley (Brookmeyer and Crowley, 1982) method.
Time Frame: Up to approximately 3 years
Population: Safety Analysis Set: all participants who were enrolled and received at least 1 dose of tarlatamab. Among the 40 participants included in the Safety Analysis Set, 35 participants died because of any cause and 5 participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tarlatamab Dose Expansion
Number analyzed (Participants) | 40
months | 7.9 [4.4 to 13.2]

8. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with a best overall response of confirmed response (CR/PR) or stable disease (SD) as per RECIST 1.1. The DCR was assessed per RECIST 1.1. The percentage of participants with disease control with corresponding exact 95% CI was calculated using the Clopper-Pearson (Clopper and Pearson, 1934) method. The result reported was evaluated by central reviewer assessment.
Time Frame: Up to approximately 3 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tarlatamab Dose Expansion
Number analyzed (Participants) | 25
percentage of participants | 36.0 [18.0 to 57.5]

9. Secondary Outcome: Maximum Serum Concentration (Cmax) of Tarlatamab
Description: Pharmacokinetic (PK) parameters of tarlatamab were determined from the time concentration profile using standard non-compartmental approaches and considering the profile over the complete sampling interval.
Time Frame: Cycle 2 Day 1 and Day 15: Predose, end of infusion (EOI), 2, 6, 24, 48, 96 and 168 hours after EOI
Population: PK Analysis Set: all participants who received at least 1 dose of tarlatamab and had at least 1 PK sample collected. The total number of participants analyzed includes only participants with available data at pre-specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Tarlatamab Dose Expansion
Number analyzed (Participants) | 25
μg/mL
  Cycle 2 Day 1 | 31.1 (26)
  Cycle 2 Day 15: number analyzed (Participants) | 21
  Cycle 2 Day 15 | 31.7 (19)

10. Secondary Outcome: Tarlatamab Concentration at the End of a Dosing Interval or Before Planned Next Dose (Ctrough)
Description: PK parameters of tarlatamab were determined from the time concentration profile using standard non-compartmental approaches and considering the profile over the complete sampling interval. The result for this endpoint is given for cycle 2 only.
Time Frame: Cycle 2 Day 15: Predose
Population: PK Analysis Set: all participants who received at least 1 dose of tarlatamab and had at least 1 PK sample collected. The number of participants analyzed only includes participants with available data for each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Tarlatamab Dose Expansion
Number analyzed (Participants) | 21
μg/mL | 5.36 (36)

11. Secondary Outcome: Area Under the Concentration-time Curve Over the Dosing Interval From Time 0 to 336 Hours (AUC336) of Tarlatamab
Description: as for outcome 10
Time Frame: Cycle 2 Day 1 and Day 15: Predose, EOI, 2, 6, 24, 48, 96, 168, and 336 hours after EOI
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Tarlatamab Dose Expansion
Number analyzed (Participants) | 25
hr*μg/mL
  Cycle 2 Day 1 | 4010 (28)
  Cycle 2 Day 15: number analyzed (Participants) | 21
  Cycle 2 Day 15 | 4260 (26)

12. Secondary Outcome: Terminal Phase Elimination Half-life (t1/2,z) of Tarlatamab
Description: as for outcome 10
Time Frame: Cycle 2 Day 15: Predose, EOI, 2, 6, 24, 48, 96 and 168 hours after EOI
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Tarlatamab Dose Expansion
Number analyzed (Participants) | 21
days | 7.23 (33)

ADVERSE EVENTS:
Time Frame: Death - From enrollment until End of Study (EOS); Median (min, max) was 6.7 (0.1, 37.4) months. TEAE - from 1st study drug until min(last dose + 65 days, EOS); Median (min, max) duration was 3.6 (1.1, 37.3) months.
Description: Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug. All-cause mortality is reported for all participants enrolled in the study.
Arm/Group | Tarlatamab Dose Expansion
All-Cause Mortality (participants affected / at risk) | 35/41
Serious Adverse Events (participants affected / at risk) | 27/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tarlatamab Dose Expansion (N=40)
Atrial flutter (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 4
Pain (General disorders) | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 1
Cytokine release syndrome (Immune system disorders) | 9
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia aspiration (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Head injury (Injury, poisoning and procedural complications) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Immobilisation syndrome (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine cancer of the prostate metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Neuroendocrine carcinoma of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Epilepsy (Nervous system disorders) | 1
Immune-mediated encephalopathy (Nervous system disorders) | 1
Neurotoxicity (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Bladder obstruction (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tarlatamab Dose Expansion (N=40)
Anaemia (Blood and lymphatic system disorders) | 14
Atrial fibrillation (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 3
Hypothyroidism (Endocrine disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 18
Diarrhoea (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 11
Asthenia (General disorders) | 4
Chills (General disorders) | 5
Fatigue (General disorders) | 16
Gait disturbance (General disorders) | 2
Malaise (General disorders) | 2
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 2
Pyrexia (General disorders) | 16
Cytokine release syndrome (Immune system disorders) | 26
COVID-19 (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 5
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 5
Blood creatine phosphokinase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 3
C-reactive protein increased (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 3
Lymphocyte count decreased (Investigations) | 3
Weight decreased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 20
Hypokalaemia (Metabolism and nutrition disorders) | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Aphasia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 17
Headache (Nervous system disorders) | 10
Neuralgia (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 5
Anxiety (Psychiatric disorders) | 4
Confusional state (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 3
Restlessness (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 4
Haematuria (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 5
Urinary retention (Renal and urinary disorders) | 7
Pelvic pain (Reproductive system and breast disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Embolism (Vascular disorders) | 2
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 4
Orthostatic hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2024-06-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT04702737/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT04702737/SAP_001.pdf